CLINICAL TRIAL: NCT01828008
Title: Treatment of CD20 Antibody Plus CIK for Patients With Refractory Lymphomas
Acronym: CIK
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Han weidong (Other)
Responsible Party: Sponsor-Investigator, Han weidong, combination of anti-CD20 with CIK for refractory lymphomas, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: BT-004
Record Dates: First submitted 2013-04-06; First posted 2013-04-10 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-01

CONDITIONS: Lymphomas
Keywords: Mabthera; cytokine induced killer cell
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To study the safety and efficacy of CD20 antibody usage followed by CIK transfusion in refractory and/or chemoresistant lymphomas.

DETAILED DESCRIPTION:
Autologous CIK transfusion within 3 days post CD20 antibody treatment.

ELIGIBILITY:
Inclusion Criteria:

- diagnosed as B-cell lymphoma with CD20 positiveness, and need to therapy

Exclusion Criteria:

- to refuse the therapy and need not tolerate the therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients with CD20-positive Lymphomas
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 5 years